CLINICAL TRIAL: NCT06613828
Title: Efficacy of Five Strategies To Improve Stroke Awareness in the Spanish-Speaking Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Juan Manuel Marquez Romero, Principal Investigator, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: F-2024-101-181
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Stroke Acute
Keywords: Stroke Symptom Recognition; Mnemonic-based education; stroke awareness; Spanish-speaking population; Public health intervention
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- RAPIDO Strategy Arm (Experimental): Participants in this arm receive educational training based on the RAPIDO strategy, an acronym developed to raise awareness of stroke symptoms among the Spanish-speaking community. This strategy is modeled after the English FAST mnemonic and focuses on the rapid identification of stroke symptoms.
  Interventions: Behavioral: Mnemonic-Based Educational Training for Stroke Symptom Recognition
- CORRE Strategy Arm (Experimental): Participants in this arm are trained using the CORRE strategy, created by a Colombian neurologist. It mirrors the structure of other mnemonic-based interventions and emphasizes the importance of quickly recognizing and acting upon early stroke symptoms.
  Interventions: Behavioral: Mnemonic-Based Educational Training for Stroke Symptom Recognition
- DALE Strategy Arm (Experimental): Participants in this arm are educated using the DALE strategy, developed in 2012 by researchers at the University of Guadalajara. Similar to the RAPIDO strategy, DALE adapts the FAST mnemonic for the Spanish-speaking population, promoting quick recognition and response to cerebrovascular symptoms.
  Interventions: Behavioral: Mnemonic-Based Educational Training for Stroke Symptom Recognition
- CAMALEON Strategy Arm (Experimental): In this arm, participants receive training based on the CAMALEON strategy, a mnemonic created in Costa Rica with the support of the pharmaceutical industry. The approach is designed to facilitate the recognition of early stroke symptoms by adapting the FAST mnemonic to Spanish.
  Interventions: Behavioral: Mnemonic-Based Educational Training for Stroke Symptom Recognition
- ICTUS 911 Strategy Arm (Experimental): Participants in this arm are educated using the ICTUS 911 strategy, which differs from the other four in that it is not directly based on a literal translation of FAST. Instead, it focuses on recognizing stroke symptoms and immediately calling emergency services (911) upon suspicion of a stroke.
  Interventions: Behavioral: Mnemonic-Based Educational Training for Stroke Symptom Recognition

INTERVENTIONS:
Behavioral: Mnemonic-Based Educational Training for Stroke Symptom Recognition — This is a Culturally Adapted Mnemonic-Based Educational Strategies for Rapid Stroke Symptom Recognition in the Spanish-Speaking Population.
  It uses five distinct mnemonic strategies (RAPIDO, CORRE, DALE, CAMALEON, ICTUS 911), each specifically tailored for a Spanish-speaking audience.
  Aims to improve the recognition of early cerebrovascular disease symptoms, differentiating it from other clinical studies that might focus on different health conditions or target populations.
  Emphasizes its focus on rapid action by educating participants about stroke symptoms and the importance of contacting emergency services (911).

SUMMARY:
The goal of this experimental study is to evaluate the efficacy of five educational strategies for recognizing early symptoms of cerebrovascular disease (CVD) in the general adult population. The main questions it aims to answer are:

- How effective are the strategies RAPIDO, CORRE, DALE, CAMALEON, and ICTUS 911 in improving the recognition of early CVD symptoms?

Researchers will compare these strategies to determine which one leads to the highest increase in symptom recognition. Participants will receive a brief educational session on one of the five strategies and will:

* Complete a pre- and post-intervention survey (Stroke Awareness Questionnaire, SAQ).
* Receive short training on CVD symptoms and the urgency of contacting emergency services.

The primary outcome is the improvement in SAQ scores, and the secondary outcome is the proportion of participants achieving adequate knowledge of CVD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age: Participants must be 18 years or older.
* Consent: Participants must provide informed consent to participate in the study.
* General Population: Participants from the general public, regardless of their health insurance status or previous medical history (except as specified in exclusion criteria).
* Language: Participants must be fluent in Spanish, as the educational interventions are based on Spanish-language mnemonic strategies.

Exclusion Criteria:

* History of Stroke: Participants with a previous diagnosis of cerebrovascular disease (stroke) will be excluded.
* Cognitive Impairment: Participants who are unable to understand or complete the Stroke Awareness Questionnaire (SAQ) due to cognitive or communication impairments will not be eligible.
* Incomplete Evaluation: Participants who are unable to complete both the pre- and post-intervention assessments will be excluded from the study.

Elimination Criteria:

* Lack of Follow-Up: Participants who fail to attend the second evaluation (7 days post-intervention) will be excluded from the final analysis.
* Withdrawal of Consent: Participants who choose to withdraw from the study at any time will be eliminated from further participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 435 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2024-11-07 (Actual)

PRIMARY OUTCOMES:
Change in Stroke Awareness Questionnaire (SAQ) Score | Pre-intervention and 7 days post-intervention.
  This measure will assess the change in participants' knowledge of stroke symptoms before and after receiving the educational intervention. The SAQ evaluates awareness of stroke symptoms, risk factors, and appropriate responses to suspected stroke events.

SECONDARY OUTCOMES:
Proportion of Participants with Adequate Knowledge of Stroke Symptoms | 7 days post-intervention.
  This outcome measures the proportion of participants who achieve a predetermined "adequate knowledge" score on the SAQ, defined as correctly identifying at least 3 stroke symptoms and understanding the need to contact emergency services (911) within 3 hours of symptom onset.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General de Zona #2, Aguascalientes, Aguascalientes, Mexico

IPD SHARING:
Plan to Share IPD: No